CLINICAL TRIAL: NCT00861276
Title: Use of Nicotine Substitute Prescribed at Hourly Intake or ad Libitum for Heavy Smokers Willing to Quit: a Randomized Controlled Trial
Brief Title: Nicotine Substitute Prescribed at Hourly Intake or ad Libitum for Heavy Smokers Willing to Quit
Acronym: SUNIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: Pharmacia (Industry)
Responsible Party: Alain Pecoud, Department of Ambulatory Care and Community Medicine, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prot 29/99
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Nicotine; Administration and dosage; Randomized Controlled Trial
MeSH Terms: conditions — Smoking Cessation | interventions — Nasal Sprays

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Arm instructed to use spray at least once an hour when awake.
  Interventions: Drug: Nasal Spray Nicotine Substitute (Experimental)
- 2 (Active Comparator): Ad libitum: patients were instructed to use NNS when craving appears.
  Interventions: Drug: Nasal Spray Nicotine Substitute (ad libitum)

INTERVENTIONS:
Drug: Nasal Spray Nicotine Substitute (Experimental) — During the first month, subjects in the intervention group received instruction from the physician to use NNS regularly (at least 2 puffs/hour, for an average of 1 mg nicotine/hour when awake).
  Other Names: Nicorette(R) nasal spray
  Arms: 1
Drug: Nasal Spray Nicotine Substitute (ad libitum) — In the control group, participants were instructed to use NNS as needed to suppress withdrawal symptoms when cravings appeared.
  Other Names: Nicorette(R) Nasal Spray
  Arms: 2

SUMMARY:
Objective: To assess the impact of instructional guidance in the regular use of use nicotine nasal spray (NNS) on the true use of NNS during the first three weeks of smoking cessation for heavy smokers who are willing to quit.

Methods: This randomized, open, controlled trial included 50 patients who were heavy smokers, were willing to quit, and attending an academic outpatient clinic in Western Switzerland. Patients were randomised to instruction on NNS use as "ad libitum" (administration whenever cravings appear; control group) or to use NNS at least every hour when awake (intervention group). Intakes were monitored using an electronic device fixed in the spray unit (MDILogTM) during the first three weeks of use. Self reported abstinence from smoking at six months was confirmed by expired-air carbon monoxide. Using intention-to-treat analysis, random-effect GLS regression was used to calculate the mean difference of daily doses between groups controlling for lack of independence between measures from the same individual.

ELIGIBILITY:
Inclusion Criteria:

* Highly dependent smokers in the stage of preparation according to Prochaska and Di Clemente's stages of change model

Exclusion Criteria:

* History of myocardial infarction in the preceding 3 months
* Pregnancy or breast-feeding
* Use of any form of smokeless tobacco or other nicotine replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2000-06; Primary Completion 2001-07 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
The daily number of intakes during the first three weeks recorded with an electronic device fixed on the spray unit (microswitch-actuated metered-dose inhaler chronology, MDILog™, model MDC-511, Medtrac, Denver, Colorado). | first 3 weeks

SECONDARY OUTCOMES:
self-reported continuous abstinence from smoking from the beginning of the substitution to the end of the 6th month of follow-up, validated by an expired-air carbon monoxide (CO) concentration of less than 10 parts per million (ppm) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Zellweger, MD, Study Director — Department of Ambulatory Care and Community Medicine, University of Lausanne
Locations (1):
- Department of Ambulatory Care and Community Medicine, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995
- [Derived] Rey L, Vaucher P, Secretan F, Zellweger JP, Bodenmann P. Use of nicotine substitute prescribed at hourly plus ab libitum intake or ad libitum for heavy smokers willing to quit: a randomized controlled trial. Subst Abuse Treat Prev Policy. 2009 Jun 2;4:12. doi: 10.1186/1747-597X-4-12. PMID 19490626